CLINICAL TRIAL: NCT04547517
Title: Psychometric Evaluation of the Traditional Chinese Version of CCS-R Practicum Evaluation and the Assessment of the Counselling Competencies Among Young Peer Counsellors in Hong Kong
Brief Title: Psychometric Evaluation of the Traditional Chinese Version of CCS-R Practicum Evaluation
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: CCS-R
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-09

CONDITIONS: Peer Group

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Evaluation of Counselling competencies — To complete a set of questionnaires

SUMMARY:
This study aims to translate the original Counselor Competencies Scale-Revised (CCS-R, English version) into traditional Chinese. It will then test the psychometric properties of the newly translated CCS-R to examine its factorial structure using both exploratory factor analysis (EFA) and CFA.

DETAILED DESCRIPTION:
Clinical supervisors are charged with facilitating the development of their supervisees toward becoming ethical and competent. In addition, clinical supervisors are expected to serve as gatekeepers for the profession and deny entry to students who demonstrate a deficiency of necessary competencies. Despite the developmental and remedial expectations for clinical supervisors, specific guidelines to direct clinical supervisors' evaluation of their supervisees' level of counseling competencies are limited. The lack of agreed-upon and standardized evaluation criteria for supervisees' minimum level of counseling competencies and the limited availability of tested assessments to measure supervisees' counseling competencies fosters subjectivity in supervisory assessment and potential remediation. Therefore, additional research is warranted relating to clinical supervisory evaluation instruments.

Supervisory evaluation is "the nucleus of clinical supervision". Specifically, "supervisors document and provide supervisees with ongoing feedback regarding their performance and schedule periodic formal evaluative sessions throughout the supervisory relationship". However, clinical supervisors are often uncomfortable in evaluating their supervisees. Nevertheless, effective and ethical supervision supports supervisees' development of counseling competencies in which supervisors provide their supervisees with both formative and summative evaluative feedback within the context of a strong supervisory alliance. Limited research was identified investigating supervisory evaluation processes with standardized assessment tools such as the counselling competencies in Hong Kong.

An initial quantitative investigation of the 23-item counselling competencies scale-revised (CCS-R) supported the construct validity (e.g., exploratory factor analysis identified a ﬁve-factor model [professional behaviors, professional behaviors, counseling skills, assessment and application, and professional dispositions], accounting for 72.61% of the variance), internal consistency reliability, interrater reliability (r ¼.570), and criterion-related validity (correlation between supervisees' practicum course grade and ﬁnal CCS score, r ¼.407,) of the instrument. The researchers concluded that "the CCS is a promising instrument for assessment in counselor education and supervision". Nevertheless, qualitative data are warranted to evaluate the CCS with a sample of clinical supervisors and their supervisees around its (a) functionality in communication of supervisory feedback with the CCS, (b) consistency in CCS evaluation, and (c) emotional reactions to supervisory evaluation with the CCS. Therefore, this study aims to translate the original Counselor Competencies Scale-Revised (CCS-R, English version) into traditional Chinese. It will then test the psychometric properties of the newly translated CCS-R to examine its factorial structure using both exploratory factor analysis (EFA) and CFA.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-35.
* Completing the training of peer counselling for smoking cessation or anti-drug abusing
* Be able to speak Cantonese and read traditional Chinese.

Exclusion Criteria:

* Those who do not provide written consent.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young people in Hong Kong who complete the training of peer counselling for smoking cessation or anti-drug abusing will be selected and invited to participate in the proposed study
Sampling Method: Non-Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Counselling Competencies | Baseline
  The counselling competencies scale-revised is a 23-item scale measuring Counselor Competencies. It includes two factors, which are counselling skills & therapeutic conditions with 12 items, and counselling dispositions &behaviors with 11 items. Each of the items has a range of 1-5 points (0 indicates poor performance, while 5 indicates performance exceeding expectations). The 12 and 11 components scores are summed to yield two scores, with a range of 12-60 points and 11-55 points respectively.

SECONDARY OUTCOMES:
Counselling performance assessment scores | Baseline
  Validated Counselling performance assessment Sheet

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Yes
The relevant anonymized patient-level data, full dataset, technical appendix, and statistical code are available on reasonable request. The approval from the Principal Investigator for the purpose of data use is required.
Supporting Information: SAP, ICF
Time Frame: After the project is completed and the results of the project have been published
Access Criteria: Request could be sent to Principal Investigator (william3@hku.hk)